CLINICAL TRIAL: NCT06306495
Title: Examination of Insomnia, Physical Activity Level and Stress Level in University Students
Brief Title: Insomnia, Physical Activity Level and Stress Level
Acronym: PA
Status: Completed | Type: Observational
Sponsor: Halic University (Other)
Responsible Party: Principal Investigator, Seda Saka, Associate Professor Doctor, Halic University
Other Study IDs: 26.01.2022/17
Record Dates: First submitted 2024-02-06; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: insomnia; physical activity; stress level
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Motor Activity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- University students: Study data will be collected with the International Physical Activity Survey, Demographic Data Form, Sleep Hygiene Index, Distress Tolerance Scale and Pittsburgh Sleep Quality Index administered to all participants.
  Interventions: Other: International Physical Activity Survey

INTERVENTIONS:
Other: International Physical Activity Survey — Study data will be collected with the International Physical Activity Survey, Demographic Data Form, Sleep Hygiene Index, Distress Tolerance Scale and Pittsburgh Sleep Quality Index administered to all participants.
  Other Names: Demographic Data Form; Sleep Hygiene Index; Distress Tolerance Scale; Pittsburgh Sleep Quality Index

SUMMARY:
Insomnia is a common, acute, intermittent, or chronic complaint of unwanted sleep difficulties characterized by sleep disturbance. Important risk factors leading to insomnia: advanced age, poor health, work stress, shift work, loss of a loved one, divorce, domestic violence, excessive anxiety, repressed personality, perfectionism, neuroticism, alcohol and substance abuse, excessive caffeine intake, excessive smoking, low socio-economic status and low physical activity level. Research shows that college students face more sleep problems than the general public. Factors that disrupt the sleep hygiene of university students; Students' excessive use of computers during lecture and exam periods, exposure to lights and screens for long periods of time, and environmental changes. The aim of this study is to determine the prevalence of insomnia in healthy individuals after the start of face-to-face education in university students after the pandemic period and to determine the physical activity associated with insomnia in this population group. Examining levels and other behavioral factors. The research was conducted on students studying at Istanbul Rumeli University, Haliç University and Yalova University between March 2022 and August 2022. It will be held online via Google Forms with students between the ages of 18-25. Study data will be collected with the International Physical Activity Survey, Demographic Data Form, Sleep Hygiene Index, Distress Tolerance Scale, and Pittsburgh Sleep Quality Index. An application will be made to obtain approval from the Haliç University Non-Interventional Clinical Research Ethics Committee. Informed consent will be obtained from people participating in the research. Statistical analysis of the data will be done with IBM SPSS 23.0 software.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-25,
* Associate and undergraduate students studying in the field of health sciences
* Agreeing to participate in the study,
* Native speaker of Turkish,
* Male and female individuals

Exclusion Criteria:

* Refusing to participate in the study,
* Having a diagnosed psychiatric illness,
* Using any medical medication that affects sleep
* Having a health condition that prevents physical activity,
* Be missing data

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population of the study is university education in the Marmara Region. consists of continuing students. The study sample consists of associate and undergraduate students studying in the field of Health Sciences, between the ages of 18-25, who continue their university education in Istanbul and Yalova.
Sampling Method: Non-Probability Sample
Enrollment: 473 (Actual)
Dates: Start 2022-03-27 (Actual); Primary Completion 2023-08-12 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Prevalence of insomnia in university students | 17 months
  It will be evaluated with the Pittsburgh Sleep Quality Index. Pittsburgh Sleep Quality Index (PSQI) is a scale that assesses sleep quality and disturbance over the past month. It consists of 24 questions, 19 of which are self-report and 5 of which are answered by a spouse or roommate. The self-report section consisting of 19 questions was used in this study. The 18 scored questions of the scale consist of 7 components (Subjective Sleep Quality, Sleep Latency, Sleep Duration, Habitual Sleep Efficiency, Sleep Disorder, Sleep Medication Use and Daytime Dysfunction). Each component is evaluated on a 0-3 point scale and the total score of the 7 components gives the total score of the scale. The total score varies between 0 and 21. A total score greater than 5 means "poor sleep quality"

SECONDARY OUTCOMES:
The effect of insomnia on physical activity level | 17 months
  It will be evaluated with the International Physical Activity Questionnaire Short Form (IPAQ-SF).IPAQ-SF was used to determine physical activity levels. This is a seven-question self-report questionnaire that assesses physical activity over the past 7 days. According to IPAQ-SF records, there are four levels of intensity: sitting, walking, moderate intensity (e.g. leisure cycling) and vigorous intensity (e.g. jogging or aerobics)
The effect of insomnia on stress levels in university students | 17 months
  It will be evaluated with the Distress Tolerance Scale (DTS).DTS; This scale aims to determine the stress endurance of the patient based on individual variations. DTS is a 15-item scale developed to measure individual differences in the capacity to withstand distress. The scale consists of 3 sub-factors (self-efficacy, tolerance, regulation). A high score on the scale indicates indicates a high level of resilience
Effects of sleep hygiene on insomnia in university students | 17 months
  Evaluated by Sleep Hygiene Index (SHI).The SHI form consists of 13 questions and evaluates the sleep behaviors that constitute the sleep hygiene of the participants. Scores ranged from 13 to 65, with higher scores indicating poorer sleep hygiene in the participants. It has been reported that participants with high scores on the form have worse sleep hygiene

CONTACTS AND LOCATIONS:
Overall Officials: Özge Ökcü, phdc, Study Director — Halic University
Locations (1):
- Halic University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sutton EL. Insomnia. Ann Intern Med. 2021 Mar;174(3):ITC33-ITC48. doi: 10.7326/AITC202103160. Epub 2021 Mar 9. PMID 33683929
- [Result] Amaral AP, Soares MJ, Pinto AM, Pereira AT, Madeira N, Bos SC, Marques M, Roque C, Macedo A. Sleep difficulties in college students: The role of stress, affect and cognitive processes. Psychiatry Res. 2018 Feb;260:331-337. doi: 10.1016/j.psychres.2017.11.072. Epub 2017 Dec 2. PMID 29227897
- [Result] Williams AB, Dzierzewski JM, Griffin SC, Lind MJ, Dick D, Rybarczyk BD. Insomnia Disorder and Behaviorally Induced Insufficient Sleep Syndrome: Prevalence and Relationship to Depression in College Students. Behav Sleep Med. 2020 Mar-Apr;18(2):275-286. doi: 10.1080/15402002.2019.1578772. Epub 2019 Feb 21. PMID 30789063
- [Result] Hartescu I, Morgan K. Regular physical activity and insomnia: An international perspective. J Sleep Res. 2019 Apr;28(2):e12745. doi: 10.1111/jsr.12745. Epub 2018 Aug 16. PMID 30117220